CLINICAL TRIAL: NCT04308161
Title: The Effectiveness of Topical Oral Vitamin D Gel in Prevention of Radiation-induced Oral Mucositis
Brief Title: Vitamin D Oral Gel for Prevention of Radiation Induced Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB NO: 00010556-IORG 0008839
Record Dates: First submitted 2020-03-12; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Oral Mucositis Due to Radiation
Keywords: vitamin D topical oral gel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vitamin D oral gel (Experimental): Topical oral vitamin D gel twice daily (Equivalent to 8000 I.U/day vitamin D) for six weeks.
  Topical oral Vitamin D gel is prepared with the aid of pharmaceutics department, faculty of pharmacy, Alexandria University. It is prepared by using Cholecalciferol 2ml ampoule (200.000 I.U.) within topical oral gel formulation.
  Interventions: Drug: vitamin D oral gel
- conventional therapy (Active Comparator): Conventional therapy (symptomatic treatment) which included:
  * Miconaz oral gel
  * BBC oral spray
  * Oracure gel
  * Alkamisr sachets
  Dose: Three times a day for six weeks
  Interventions: Drug: Miconazole Topical Gel; Drug: BBC oral spray; Drug: Oracure gel; Other: Alkamisr sachets
- combination therapy (Experimental): Topical oral vitamin D gel twice daily (Equivalent to 8000 I.U/day vitamin D) for six weeks in combination with the symptomatic treatment
  Symptomatic treatment which included:
  * Miconaz oral gel
  * BBC oral spray
  * Oracure gel
  * Alkamisr sachets
  Symptomatic treatment dose: Three times a day for six weeks
  Interventions: Drug: vitamin D oral gel; Drug: Miconazole Topical Gel; Drug: BBC oral spray; Drug: Oracure gel; Other: Alkamisr sachets

INTERVENTIONS:
Drug: vitamin D oral gel — vitamin D is a fat soluble vitamin which has important calcemic roles in the body regarding bone homeostasis and calcium/phosphorus balance. Recently, the non-calcemic roles of vitamin D as anti-inflammatory, anti-oxidant and immuno-regulatory functions have been widely reported.So, we tried to use it for prevention of radiation induced oral mucositis
  Arms: combination therapy; vitamin D oral gel
Drug: Miconazole Topical Gel — topical anti fungal agent
  Arms: combination therapy; conventional therapy
Drug: BBC oral spray — Topical anesthetics and anti-inflammatory agent
  Arms: combination therapy; conventional therapy
Drug: Oracure gel — Topical analgesic gel
  Arms: combination therapy; conventional therapy
Other: Alkamisr sachets — Sodium bicarbonate mouthwash
  Arms: combination therapy; conventional therapy

SUMMARY:
The main aim of this study was to evaluate clinically the effect of topical oral vitamin D gel in comparison to conventional therapy in prevention of radiation - induced oral mucositis

DETAILED DESCRIPTION:
The study was designed as randomized, controlled, clinical trial. patients who were undergoing to receive radiotherapy were divided into three groups: Group I: was given conventional treatment.Group II : was given topical oral gel of vitamin D. Group III: was given topical oral gel of vitamin D in combination with the conventional treatment.

All patients were clinically evaluated at the start the radiotherapy, three weeks and six weeks later for pain and oral mucositis severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to receive radiotherapy as a treatment of head and neck cancer either as postoperative (adjuvant) therapy or definitive therapy.
* Patients whose radiotherapy treatment planned dose is 50 Gy or above.
* Patients receiving radiotherapy alone or receiving concomitant cisplatin (or carboplatin) with radiotherapy.

Exclusion Criteria:

* Patients under Anticoagulants such as warfarin, heparin, or aspirin.
* Patients whose radiotherapy treatment planned dose is lower than 50 Gy.
* Patients suffering from any uncontrolled systemic diseases (such as diabetes, cardiovascular, liver disorder, renal dysfunction)
* Patients with findings of any physical or mental abnormality which would interfere with or be affected by the study procedure.
* Hyper-calcemic patients.
* Smokers.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in severity of oral mucositis at different time points along the study | up to 3 and 6 weeks
  Oral mucositis will be evaluated by the World Health Organization (WHO) scale which record the extent and severity of oral mucositis at the third and sixth week after the first radiotherapy session.

SECONDARY OUTCOMES:
Pain and discomfort severity at different time points along the study: Numeric Rating Scale | up to 3 and 6 weeks
  Discomfort and pain severity were reported by each patient using Numeric Rating Scale (NRS) at the third and sixth week after the first radiotherapy session.

CONTACTS AND LOCATIONS:
Overall Officials: Islam s Bakr, BDS, Principal Investigator — Alexandria University; azza m zaki, Phd, Study Director — Alexandria University; Riham m El-Moslemany, Phd, Study Director — Alexandria University; Rasha o Elsaka, Phd, Study Director — Alexandria University
Locations (1):
- Outpatient clinic of Department of Clinical Oncology, Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muanza TM, Cotrim AP, McAuliffe M, Sowers AL, Baum BJ, Cook JA, Feldchtein F, Amazeen P, Coleman CN, Mitchell JB. Evaluation of radiation-induced oral mucositis by optical coherence tomography. Clin Cancer Res. 2005 Jul 15;11(14):5121-7. doi: 10.1158/1078-0432.CCR-05-0403. PMID 16033826
- [Background] Maria OM, Eliopoulos N, Muanza T. Radiation-Induced Oral Mucositis. Front Oncol. 2017 May 22;7:89. doi: 10.3389/fonc.2017.00089. eCollection 2017. PMID 28589080
- [Background] Rogulj AA, Brzak BL, Boras VV, Brailo V, Milenović M. Oral complications of head and neck irradiation. Libr Oncol. 2017;45(2-3):89-93.
- [Background] Barkokebas A, Silva IH, de Andrade SC, Carvalho AA, Gueiros LA, Paiva SM, Leao JC. Impact of oral mucositis on oral-health-related quality of life of patients diagnosed with cancer. J Oral Pathol Med. 2015 Oct;44(9):746-51. doi: 10.1111/jop.12282. Epub 2014 Oct 25. PMID 25345344
- [Background] Duncan GG, Epstein JB, Tu D, El Sayed S, Bezjak A, Ottaway J, Pater J; National Cancer Institute of Canada Clinical Trials Group. Quality of life, mucositis, and xerostomia from radiotherapy for head and neck cancers: a report from the NCIC CTG HN2 randomized trial of an antimicrobial lozenge to prevent mucositis. Head Neck. 2005 May;27(5):421-8. doi: 10.1002/hed.20162. PMID 15782422
- [Background] Georgiou M, Patapatiou G, Domoxoudis S, Pistevou-Gompaki K, Papanikolaou A. Oral Mucositis: understanding the pathology and management. Hippokratia. 2012 Jul;16(3):215-6. PMID 23935285
- [Background] Sonis ST. Oral mucositis in cancer therapy. J Support Oncol. 2004 Nov-Dec;2(6 Suppl 3):3-8. PMID 15605918
- [Background] Lee CS, Ryan EJ, Doherty GA. Gastro-intestinal toxicity of chemotherapeutics in colorectal cancer: the role of inflammation. World J Gastroenterol. 2014 Apr 14;20(14):3751-61. doi: 10.3748/wjg.v20.i14.3751. PMID 24744571
- [Background] Volpato LE, Silva TC, Oliveira TM, Sakai VT, Machado MA. Radiation therapy and chemotherapy-induced oral mucositis. Braz J Otorhinolaryngol. 2007 Jul-Aug;73(4):562-8. doi: 10.1016/s1808-8694(15)30110-5. PMID 17923929
- [Background] Elad S, Zadik Y. Chronic oral mucositis after radiotherapy to the head and neck: a new insight. Support Care Cancer. 2016 Nov;24(11):4825-30. doi: 10.1007/s00520-016-3337-5. Epub 2016 Jul 30. PMID 27475958
- [Background] Wuketich S, Hienz SA, Marosi C. Prevalence of clinically relevant oral mucositis in outpatients receiving myelosuppressive chemotherapy for solid tumors. Support Care Cancer. 2012 Jan;20(1):175-83. doi: 10.1007/s00520-011-1107-y. Epub 2011 Feb 18. PMID 21331484
- [Background] Peppone LJ, Mustian KM, Morrow GR, Dozier AM, Ossip DJ, Janelsins MC, Sprod LK, McIntosh S. The effect of cigarette smoking on cancer treatment-related side effects. Oncologist. 2011;16(12):1784-92. doi: 10.1634/theoncologist.2011-0169. Epub 2011 Dec 1. PMID 22135122
- [Background] Alongi F, Giaj-Levra N, Sciascia S, Fozza A, Fersino S, Fiorentino A, Mazzola R, Ricchetti F, Buglione M, Buonfrate D, Roccatello D, Ricardi U, Bisoffi Z. Radiotherapy in patients with HIV: current issues and review of the literature. Lancet Oncol. 2017 Jul;18(7):e379-e393. doi: 10.1016/S1470-2045(17)30440-0. PMID 28677574
- [Background] Villa A, Sonis ST. Mucositis: pathobiology and management. Curr Opin Oncol. 2015 May;27(3):159-64. doi: 10.1097/CCO.0000000000000180. PMID 25774860
- [Background] Herrstedt J. Prevention and management of mucositis in patients with cancer. Int J Antimicrob Agents. 2000 Oct;16(2):161-3. doi: 10.1016/s0924-8579(00)00232-6. PMID 11053801
- [Background] Tsujimoto T, Yamamoto Y, Wasa M, Takenaka Y, Nakahara S, Takagi T, Tsugane M, Hayashi N, Maeda K, Inohara H, Uejima E, Ito T. L-glutamine decreases the severity of mucositis induced by chemoradiotherapy in patients with locally advanced head and neck cancer: a double-blind, randomized, placebo-controlled trial. Oncol Rep. 2015 Jan;33(1):33-9. doi: 10.3892/or.2014.3564. Epub 2014 Oct 23. PMID 25351453
- [Background] Wink K, Brett W. [Alcoholic cardiomyopathy]. Med Monatsschr. 1976 Nov;30(11):485-9. No abstract available. German. PMID 136590
- [Background] Patni N, Patni S, Bapna A. The optimal use of granulocyte macrophage colony stimulating factor in radiation induced mucositis in head and neck squamous cell carcinoma. J Cancer Res Ther. 2005 Jul-Sep;1(3):136-41. doi: 10.4103/0973-1482.19589. PMID 17998644
- [Background] Lalla RV, Sonis ST, Peterson DE. Management of oral mucositis in patients who have cancer. Dent Clin North Am. 2008 Jan;52(1):61-77, viii. doi: 10.1016/j.cden.2007.10.002. PMID 18154865
- [Background] Cirillo N, Vicidomini A, McCullough M, Gambardella A, Hassona Y, Prime SS, Colella G. A hyaluronic acid-based compound inhibits fibroblast senescence induced by oxidative stress in vitro and prevents oral mucositis in vivo. J Cell Physiol. 2015 Jul;230(7):1421-9. doi: 10.1002/jcp.24908. PMID 25536474
- [Background] Moslehi A, Taghizadeh-Ghehi M, Gholami K, Hadjibabaie M, Jahangard-Rafsanjani Z, Sarayani A, Javadi M, Esfandbod M, Ghavamzadeh A. N-acetyl cysteine for prevention of oral mucositis in hematopoietic SCT: a double-blind, randomized, placebo-controlled trial. Bone Marrow Transplant. 2014 Jun;49(6):818-23. doi: 10.1038/bmt.2014.34. Epub 2014 Mar 10. PMID 24614837
- [Background] Jadaud E, Bensadoun R. Low-level laser therapy: a standard of supportive care for cancer therapy-induced oral mucositis in head and neck cancer patients? Laser Ther. 2012 Dec 26;21(4):297-303. doi: 10.5978/islsm.12-RE-01. PMID 24511199
- [Background] Abdel Moneim AE, Guerra-Librero A, Florido J, Shen YQ, Fernandez-Gil B, Acuna-Castroviejo D, Escames G. Oral Mucositis: Melatonin Gel an Effective New Treatment. Int J Mol Sci. 2017 May 7;18(5):1003. doi: 10.3390/ijms18051003. PMID 28481279
- [Background] Spielberger R, Stiff P, Bensinger W, Gentile T, Weisdorf D, Kewalramani T, Shea T, Yanovich S, Hansen K, Noga S, McCarty J, LeMaistre CF, Sung EC, Blazar BR, Elhardt D, Chen MG, Emmanouilides C. Palifermin for oral mucositis after intensive therapy for hematologic cancers. N Engl J Med. 2004 Dec 16;351(25):2590-8. doi: 10.1056/NEJMoa040125. PMID 15602019
- [Background] Nair R, Maseeh A. Vitamin D: The "sunshine" vitamin. J Pharmacol Pharmacother. 2012 Apr;3(2):118-26. doi: 10.4103/0976-500X.95506. PMID 22629085
- [Background] Albahrani AA, Greaves RF. Fat-Soluble Vitamins: Clinical Indications and Current Challenges for Chromatographic Measurement. Clin Biochem Rev. 2016 Feb;37(1):27-47. PMID 27057076
- [Background] Sardar S, Chakraborty A, Chatterjee M. Comparative effectiveness of vitamin D3 and dietary vitamin E on peroxidation of lipids and enzymes of the hepatic antioxidant system in Sprague--Dawley rats. Int J Vitam Nutr Res. 1996;66(1):39-45. PMID 8698545
- [Background] Adeeb F, Khan MU, Li X, Stack AG, Devlin J, Fraser AD. High Vitamin D Levels May Downregulate Inflammation in Patients with Behcet's Disease. Int J Inflam. 2017;2017:8608716. doi: 10.1155/2017/8608716. Epub 2017 Jun 4. PMID 28660088
- [Background] Hassanalilou T, Khalili L, Ghavamzadeh S, Shokri A, Payahoo L, Bishak YK. Role of vitamin D deficiency in systemic lupus erythematosus incidence and aggravation. Auto Immun Highlights. 2017 Dec 26;9(1):1. doi: 10.1007/s13317-017-0101-x. PMID 29280010
- [Background] Abbas S, Linseisen J, Slanger T, Kropp S, Mutschelknauss EJ, Flesch-Janys D, Chang-Claude J. Serum 25-hydroxyvitamin D and risk of post-menopausal breast cancer--results of a large case-control study. Carcinogenesis. 2008 Jan;29(1):93-9. doi: 10.1093/carcin/bgm240. Epub 2007 Oct 31. PMID 17974532
- [Background] Ng K, Meyerhardt JA, Wu K, Feskanich D, Hollis BW, Giovannucci EL, Fuchs CS. Circulating 25-hydroxyvitamin d levels and survival in patients with colorectal cancer. J Clin Oncol. 2008 Jun 20;26(18):2984-91. doi: 10.1200/JCO.2007.15.1027. PMID 18565885
- [Background] Tretli S, Hernes E, Berg JP, Hestvik UE, Robsahm TE. Association between serum 25(OH)D and death from prostate cancer. Br J Cancer. 2009 Feb 10;100(3):450-4. doi: 10.1038/sj.bjc.6604865. Epub 2009 Jan 20. PMID 19156140
- [Background] Mokhtari Z, Hekmatdoost A, Nourian M. Antioxidant efficacy of vitamin D. J Parathyr Dis [Internet]. 2016;5(1):11-6.
- [Background] Barragan M, Good M, Kolls JK. Regulation of Dendritic Cell Function by Vitamin D. Nutrients. 2015 Sep 21;7(9):8127-51. doi: 10.3390/nu7095383. PMID 26402698
- [Background] Calton EK, Keane KN, Newsholme P, Soares MJ. The Impact of Vitamin D Levels on Inflammatory Status: A Systematic Review of Immune Cell Studies. PLoS One. 2015 Nov 3;10(11):e0141770. doi: 10.1371/journal.pone.0141770. eCollection 2015. PMID 26528817
- [Background] Oosterom N, Dirks NF, Heil SG, de Jonge R, Tissing WJE, Pieters R, van den Heuvel-Eibrink MM, Heijboer AC, Pluijm SMF. A decrease in vitamin D levels is associated with methotrexate-induced oral mucositis in children with acute lymphoblastic leukemia. Support Care Cancer. 2019 Jan;27(1):183-190. doi: 10.1007/s00520-018-4312-0. Epub 2018 Jun 19. PMID 29922939
- [Background] Christopher I, Ramsey P, Chant GR, Lockley AR, Gb W, Fields B, et al. ( 12 ) United States Patent ( 10 ) Patent No .: 2015;2(12).
- [Background] Anand A, Singh S, Sonkar AA, Husain N, Singh KR, Singh S, Kushwaha JK. Expression of vitamin D receptor and vitamin D status in patients with oral neoplasms and effect of vitamin D supplementation on quality of life in advanced cancer treatment. Contemp Oncol (Pozn). 2017;21(2):145-151. doi: 10.5114/wo.2017.68623. Epub 2017 Jun 30. PMID 28947884
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Killeen PR. An alternative to null-hypothesis significance tests. Psychol Sci. 2005 May;16(5):345-53. doi: 10.1111/j.0956-7976.2005.01538.x. PMID 15869691
- [Background] Daniel W. Biostatistics. A foundation for analysis in the health science. 6th edition, NewYork: John Wiley and sons, Inc; 1995.
- [Background] Pannucci CJ, Wilkins EG. Identifying and avoiding bias in research. Plast Reconstr Surg. 2010 Aug;126(2):619-625. doi: 10.1097/PRS.0b013e3181de24bc. PMID 20679844
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Musha A, Shimada H, Shirai K, Saitoh J, Yokoo S, Chikamatsu K, Ohno T, Nakano T. Prediction of Acute Radiation Mucositis using an Oral Mucosal Dose Surface Model in Carbon Ion Radiotherapy for Head and Neck Tumors. PLoS One. 2015 Oct 29;10(10):e0141734. doi: 10.1371/journal.pone.0141734. eCollection 2015. PMID 26512725
- [Background] McGuire DB, Correa ME, Johnson J, Wienandts P. The role of basic oral care and good clinical practice principles in the management of oral mucositis. Support Care Cancer. 2006 Jun;14(6):541-7. doi: 10.1007/s00520-006-0051-8. Epub 2006 Apr 25. PMID 16775649
- [Background] Vashi PG, Trukova K, Lammersfeld CA, Braun DP, Gupta D. Impact of oral vitamin D supplementation on serum 25-hydroxyvitamin D levels in oncology. Nutr J. 2010 Nov 23;9:60. doi: 10.1186/1475-2891-9-60. PMID 21092237
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045